CLINICAL TRIAL: NCT05916729
Title: "The Effect of Using Preparations With Maqui Berry Extract in Treating Oral Candidiasis in Patients With Diabetes Mellitus and Systemically Healthy Persons"
Brief Title: Use of Maqui Berry Extract in Treating Oral Candidiasis in Diabetes Mellitus Patients and Systemically Healthy Persons
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Natasa Nikolic Jakoba, Assist. Prof., University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBelgrade 36/9
Record Dates: First submitted 2023-06-11; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Oral Candidiases
MeSH Terms: conditions — Candidiasis, Oral | interventions — Miconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Healthy subjects with acrylate dentures and oral Candida spp infection-Miconazole group (Active Comparator): These group includes systematically healthy patients wearing acrylate dentures and with microbiologically confirmed oral infection caused with Candida spp.
  These patients were treated with Miconazole gel.
  Interventions: Drug: Miconazole
- Healthy subjects with acrylate dentures and oral Candida spp infection-Candberrol-Miconazole group (Experimental): These group includes systematically healthy patients wearing acrylate dentures and with microbiologically confirmed oral infection caused with Candida spp.
  These patients were treated with Miconazole gel and Candberrol lozenges.
  Interventions: Drug: Miconazole; Dietary Supplement: CandBerrol® lozenges
- Diabetic subjects without dentures and with oral Candida spp infection - Miconazole group (Active Comparator): These group includes diabetes mellitus patients without acrylate dentures and with microbiologically confirmed oral infection caused with Candida spp.
  These patients were treated with Miconazole gel.
  Interventions: Drug: Miconazole
- Diabetic subjects without dentures and with oral Candida spp infection - Miconazole-Candberrol group (Experimental): These group includes diabetes mellitus patients without acrylate dentures and with microbiologically confirmed oral infection caused with Candida spp.
  These patients were treated with Miconazole gel and Candberrol lozenges.
  Interventions: Drug: Miconazole; Dietary Supplement: CandBerrol® lozenges
- Diabetic subjects with acrylate dentures and oral Candida spp - Miconazole group (Active Comparator): These group includes diabetes mellitus patients with acrylate dentures and microbiologically confirmed oral infection caused with Candida spp.
  These patients were treated with Miconazole gel.
  Interventions: Drug: Miconazole
- Diabetic subjects with acrylate dentures and oral Candida spp - Miconazole and Candberrol group (Experimental): These group includes diabetes mellitus patients with acrylate dentures and microbiologically confirmed oral infection caused with Candida spp.
  These patients were treated with Miconazole gel and Candberrol lozenges.
  Interventions: Drug: Miconazole; Dietary Supplement: CandBerrol® lozenges

INTERVENTIONS:
Drug: Miconazole — Protocol for active control groups includes use of Miconazole Oral gel for 14 days with frequency of four time per day.
  Other Names: Daktanol®
Dietary Supplement: CandBerrol® lozenges — Protocol for experimental groups includes use of Miconazole Oral gel and CandBerrol® lozenges for 14 days with frequency of four time per day
  Arms: Diabetic subjects with acrylate dentures and oral Candida spp - Miconazole and Candberrol group; Diabetic subjects without dentures and with oral Candida spp infection - Miconazole-Candberrol group; Healthy subjects with acrylate dentures and oral Candida spp infection-Candberrol-Miconazole group

SUMMARY:
Fungi from the genus Candida present the saprophytic flora of the cavity. This saprophytic yeast can cause different form of oral infections at immunocompromised patients as well as at subjects with impaired local oral microbiota e.g. wearers of dentures.

The most common cause of oral candidiasis is Candida albicans, but recently, non-albicans species has also been commonly isolated. One of the reasons for growing frequency of non-albicans species is traditional antifungal therapy. Standard antifungal therapy, which means elimination of yeasts, lead to antimicrobial resistance, dysbiosis and higher incidence of non-albicans species In order to overcome these limitations, the new antimicrobial therapy is based on anti-virulence strategy. This approach relays on disarming the microorganism, instead of killing or stopping their growth, which is especially important for saprophytes.

In case of Candida albicans the main goal is preventing transition from cell to hyphal form.

DETAILED DESCRIPTION:
The aim of this study is to assess the efficiency of a dietary supplement based on Maqui Berry extract (CandBerrol® lozenge, Phytonet, Serbia) in treatment of oral candidiasis in patients who are treated with standard antifungal therapy - miconazole, 2%, (Daktanol® oral gel, Galenika, Serbia).

The study would be conducted at Clinic for Periodontology and Oral Medicine, School of Dental Medicine, University of Belgrade. The subjects would be recruited from the pool of patients who come for the treatment of suspected oral candidiasis.

A total of 90 patients with confirmed fungal infection (Candida spp.) of the oral cavity would be included in the study and divided into three groups (30 subjects per group), matched by gender and age:

Group A: systemically healthy subjects wearing acrylate dentures

Group B: subjects with diabetes mellitus without acrylate dentures

Group C: subjects with diabetes mellitus wearing acrylate dentures

Each group is further subdivided into two treatment subgroups:

1. Active control, treated with miconazole, 2% (Daktanol® oral gel, Galenika, Serbia).
2. Experimental, treated with miconazole, 2% with Maqui Berry extract (CandBerrol® lozenge, Phytonet, Serbia)

During the first examination, patients signed their consent to participate in the research based on written and oral information about the type, duration and expected outcome of the research. Following signing the consent, the research sheet specifically designed for this study would be fulfilled.

Both therapy protocol (active control and experimental therapy) would be administrated for 14 days. Therapy protocols would also include advices for oral and denture hygiene and diet. Clinical and microbiological controls would be conducted after 7th, 18th and 30th days from the start of therapy.

Patients who would not be able to follow the study instructions, would be excluded from the study.

Statistical analysis would be analyzed using the SPSS software program using appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Candida spp. infection (Clinical signs, symptoms and microbiological confirmation of infection)
* Systematically healthy wearing acrylate denture (Group A)
* Diabetic patients with/without acrylate denture (Groups B and C)

Exclusion Criteria:

* Presence of other systemic diseases
* Presence other oral mucosal contions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Presence of Candida albicans after therapy at first reexamination | 1.5 year
  Evaluation of symptoms and the presence of Candida spp. on day 18 from the beginning of the therapy
Presence of Candida albicans after therapy at second reexamination | 1.5 year
  Evaluation of symptoms and the presence of Candida spp. on day 30 from the beginning of the therapy
Presence of Candida albicans after therapy at third reexamination | 1.5 year
  Evaluation of symptoms and the presence of Candida spp. 4 days after the end of the therapy
Presence of Candida albicans after therapy at fourth reexamination | 1.5 year
  Evaluation of symptoms and the presence of Candida spp. 12 days after the end of the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Natasa Nikolic Jakoba, Principal Investigator — University of Belgrade, School of Dental Medicine, Department of Periodontology
Locations (1):
- Natasa Nikolic Jakoba, Belgrade, Serbia